CLINICAL TRIAL: NCT02377960
Title: Check and Support -Pragmatic Randomized Controlled Study of the Effectiveness of 12 Month SMS-Text Message Support and IMB-based Initiation of Medication in Adults With Hypertension for Better Blood Pressure Control and Medication Adherence
Brief Title: Check and Support -Enhancing the Treatment of Hypertension in Outpatient Care, a Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Health Centre of Jyväskylä Cooperation Area (Unknown); Central Finland Hospital District (Other); Occupational Health Care Työterveys Aalto (Unknown); Mehiläinen Jyväskylä Occupational health services (Unknown); Northern Savo Hospital District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KUH500SH01
Record Dates: First submitted 2015-01-15; First posted 2015-03-04 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Hypertension; Blood Pressure; Patient Compliance; Patient Adherence; Medication Adherence
Keywords: SMS; text message; mHealth; IMB
MeSH Terms: conditions — Hypertension; Patient Compliance; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (Reference group) (Active Comparator): Treatment is leaded by treating physician according to national guide lines with no study-specific medication or clinical appointment protocol.
  Interventions: Behavioral: Usual care
- An IMB model-based initiation of medication (Experimental): In addition to usual care, participants allocated to intervention group will receive
  An IMB model-based initiation of medication i.e. a nine-point check list to be fulfilled by physician and patient together when ordering the antihypertensive medication for the first time
  Interventions: Behavioral: IMB model-based initiation of antihypertensive medication; Behavioral: Tailored SMS-text message support
- Tailored SMS-text message support (Experimental): Tailored SMS-text message support for the first 12 months of medication. At the beginning (2 weeks), text messages are send on daily basis and focused on medications-reminders and coping with potential side-effects of medication.
  After that, text messages will be sent less often and the focus will change to keeping up with medication and reminding of importance of performing adequate home BP self-monitoring, achieving the BP target and attending clinical appointments.
  Interventions: Behavioral: IMB model-based initiation of antihypertensive medication; Behavioral: Tailored SMS-text message support

INTERVENTIONS:
Behavioral: IMB model-based initiation of antihypertensive medication — 1.An IMB model-based initiation of medication i.e. a nine-point check list to be fulfilled by physician and patient together when ordering the antihypertensive medication for the first time
  Other Names: Check list for initiation of antihypertensive medication
  Arms: An IMB model-based initiation of medication; Tailored SMS-text message support
Behavioral: Tailored SMS-text message support — 2.Tailored SMS-text message support for the first 12 months of medication. At the beginning (2 weeks), text messages are send on daily basis and focused on medications-reminders and coping with potential side-effects of medication. After that, text messages will be sent less often and the focus will change to keeping up with medication and reminding of importance of performing adequate home BP self-monitoring, achieving the BP target and attending clinical appointments.
  Other Names: Text message support
  Arms: An IMB model-based initiation of medication; Tailored SMS-text message support
Behavioral: Usual care — Usual care
  Other Names: Standard care
  Arms: Usual care (Reference group)

SUMMARY:
The purpose of this pragmatic multi-centre, cluster randomized controlled trial is to test the effectiveness of tailored SMS-text message support combined with an information-motivation-behavioral skills (IMB) model-based initiation of medication in helping outpatient care patients with hypertension to achieve blood pressure target and to enhance medication adherence.

DETAILED DESCRIPTION:
Background

Usual blood pressure is strongly related to vascular and overall mortality and high blood pressure is globally the leading risk factor for cardiovascular and related diseases. It is also well established that pharmacologic blood pressure reduction prevents cardiovascular events and deaths in persons with hypertension.

Today's physicians have plenty of knowledge and multiple effective and safety tools to treat hypertension but still majority of patients with antihypertensive medication do not achieve the blood pressure target. Poor medication adherence has been widely accepted to be the most important factor in failing to control hypertension and even 50% of hypertensive patients quit the antihypertensive medication during the first year of medication.

Numerous interventions to enhance medication adherence have been developed but even though, an intervention effective, simple and low cost enough to be carried out wide-scale in non-research settings is still to be found.

Objectives

To test whether a tailored SMS-text message support combined with an IMB model-based initiation of medication will increase the proportion of patients achieving the systolic blood pressure target at 12-month follow-up compared to usual care.

Additional objectives include investigating whether the intervention have effect on

* Medication adherence
* Systolic and diastolic blood pressure level
* Hypertension-related use of health care services
* Blood glucose, blood cholesterol, microalbuminuria, creatinine, ECG, body mass index, waist circumference exercising habits, smoking and alcohol use
* Perceived quality of life at base line and at 12-month follow-up
* Setting (physicians) and knowing (participants) an adequate BP target

And, besides

Detecting the participants who especially benefit from intervention

* Analyzing the quality and quantity of self-monitored BP and
* Assessing whether the IMB model-based structured initiation of medication can be used for screening of non-compliant patients and directing resources more accurately to them
* Collecting and analyzing participants' and physicians' feedback for future development of intervention

Study design

Pragmatic randomized controlled multicenter trial. The eight study centers are grouped to comparable pairs and randomized to function as intervention and control sites (2-cluster design).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of hypertension
* About to start medication for hypertension for the first time
* Aged 30-75 years
* Must own a mobile phone
* Must be able to read text messages
* Must be able to master own medication
* Must be able to perform home BP measurements
* Must agree in using electric drug prescription (standard in Finnish health care)

Exclusion Criteria:

* Having or is suspected to have depression or psychosis
* Serious disease, which is evaluated to have an impact on life expectancy
* Atrial flutter or atrial fibrillation
* Previous history of antihypertensive medication
* Pregnancy
* Not willing to give informed consent and take part in the study
* Systolic BP more than 200 mmHg
* Diastolic BP more than 120 mmHg
* Sudden onset or worsening of hypertension
* Clinical signs of kidney disease: proteinuria (du-prot > 500 mg), glomerulus filtration rate (eGFR) less than 45 ml/min or hypokalemia

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving the systolic blood pressure target at 12-month follow-up | 12 months from baseline
  The proportion of patients (%) achieving systolic office blood pressure (BP) target (<140 mmHg) and home BP target (<135 mmHg) are both analyzed separately using mixed effects model.
  Both office BP and home BP are measured with a validated blood pressure monitoring device (Microlife Watch BP Home A or Microlife Watch BP Home N) after appropriate rest from the left arm with an appropriately sized semi-rigid conical cuff. Office BP is the mean of three measurements separated by 15 seconds. Home BP is measured correspondingly three times in the morning and in the evening on 7 consecutive days at 12 months. Home BP is the mean of all available measurements.

SECONDARY OUTCOMES:
Measured medication adherence | 12 months from baseline
  Medication adherence is assessed by pharmacy refill data and by self-report strategy (Morisky Medication Adherence Scale, MMAS-8). Tresholds for good adherence are correspondingly (i) Medication possession ratio (MPR) 80 % or more and (ii) MMAS-8 with a score of 6 or more. Both are analyzed separately using generalized mixed effects model.
  Besides, medication adherence is analyzed as follows:
  * Persistence: time (days) from the newly initiated medication order to (i) last dispensation before failing to refill within 180 days or (ii) end of follow-up period
  * Early non-persistence: newly initiated medication order dispensed within 30 days of the initial order with no refills within 180 days
  * Primary non-adherence: newly initiated medication order not dispensed within 30 days of the initial order
Change in systolic and diastolic blood pressure | 12 months from baseline
  Both office BP and home BP are measured with a validated blood pressure monitoring device (Microlife Watch BP Home A or Microlife Watch BP Home N) after appropriate rest from the left arm with an appropriately sized semi-rigid conical cuff. Office BP is the mean of three measurements separated by 15 seconds. Home BP is measured correspondingly three times in the morning and evening on 7 consecutive days at 12 months. Home BP is the mean of all available measurements.
  Change in office BP and home BP are both analyzed separately using generalized mixed effects model. Change in systolic and diastolic blood pressure are as well both analyzed separately using generalized mixed effects model.
Hypertension-related use of health care services | 0-12 months from baseline
  Hypertension-related use of health care services (outpatient care and hospital admissions) is assessed by examining participants' electronic health records and with a questionnaire regarding the use of health services other than study centers. Proportion of scheduled clinic appointments attended is also analyzed.
Perceived quality of life | baseline and 12 months from baseline
  Perceived quality of life is assessed by EQ-5D-5L questionnaire
The proportion of participants knowing the adequate home BP target | baseline and 12 months from baseline
  Knowing the target is assessed by questionnaire at baseline and at 12 months. The results are divided into three groups: (i) knows the adequate target (ii) knows the target but it is not adequate (iii) do not know the target.
  The target is considered adequate if it differs less than 5/3 mmHg from the Finnish national guide lines for treating hypertension (Office BP target <140/90 mmHg except diabetics <140/80 mmHg. Home BP target <135/85 mmHg except diabetics <135/75 mmHg)
The proportion of patients whose BP target is adequately set | 12 months from baseline
  Setting the target is assessed by examining the electric health record at 12 months The results are divided into three groups: (i) written target is set and adequate (ii) written target is set but not adequate and (iii) written target is not set.
  The target is considered adequate if it differs less than 5/3 mmHg from the national guide lines for treating hypertension (Office BP target <140/90 mmHg except diabetics <140/80 mmHg. Home BP target <135/85 mmHg except diabetics <135/75 mmHg)
The quality and quantity of self-monitored blood pressure | baseline and 12 months from baseline
  The quality and quantity of self-monitored blood pressure measurements made prior to follow-up period is assessed first at base line. All participants are then equipped with a validated blood pressure monitoring device (Microlife Watch BP Home A or Microlife Watch BP Home N) with a memory space up to 250 measurements. The quality and quantity of self-monitored blood pressure measurements during the follow-up is assessed by examining the memory of every single device at and,the written follow-up form filled up by each participant at 12 months.
  The target is considered adequate if it differs less than 5/3 mmHg from the national guide lines for treating hypertension (Office BP target <140/90 mmHg except diabetics <140/80 mmHg. Home BP target <135/85 mmHg except diabetics <135/75 mmHg)
ECG | baseline and 12 months from baseline
  ECG is taken at baseline (timeframe 6 months before - 1 month after initiation of medication) and at 12 months.
Blood glucose level | baseline and 12 months from baseline
  Blood glucose level is tested at baseline (timeframe 6 months before - 1 month after initiation of medication) and at 12 months.
Blood cholesterol level | baseline and 12 months from baseline
  Blood cholesterol level is tested at baseline (timeframe 6 months before - 1 month after initiation of medication) and at 12 months.
Microalbuminuria | baseline and 12 months from baseline
  The presence of microalbuminuria is tested at baseline (timeframe 6 months before - 1 month after initiation of medication) and at 12 months.
Creatinine level | baseline and 12 months from baseline
  Creatinine level is tested at baseline (timeframe 6 months before - 1 month after initiation of medication) and at 12 months.
Body mass index | baseline and 12 months from baseline
  Participant's height and weight are measured by nurse/treating physician and BMI calculated at baseline and at 12 month.
Waist circumference | baseline and 12 months from baseline
  Participant's waist circumference is measured by nurse/treating physician at baseline and at 12 month.
Exercising habits | baseline and 12 months from baseline
  Every participant meets a query measuring participants' exercising habits (Kasari -index) at baseline and at 12 months.
Smoking | baseline and 12 months from baseline
  Every participant meets a query measuring participants' smoking (Heaviness of smoking -index) at baseline and at 12 months.
Alcohol use | baseline and 12 months from baseline
  Every participant meets a query measuring participants' alcohol use (Audit-c) at baseline and at 12 months.

OTHER OUTCOMES:
The quality of IMB model-based structured initiation of medication for screening of non-compliant patients | 12 months from baseline
  IMB model-based initiation of medication (check list for the initiation) includes a 10-grade numeric rating scale asking the participant to evaluate the necessity of antihypertensive medication at individual level. Our hypothesis is that the evaluated necessity of antihypertensive medication is related to medication adherence and achieving blood pressure target.

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Mäntyselkä, MD,Prof., Study Chair — University of Eastern Finland; Aapo Tahkola, LM,PHD st., Principal Investigator — Health Centre of Jyväskylä Cooperation Area
Locations (6):
- Finland (6):
  - Health Centre of Jyväskylä Cooperation Area, Jyväskylä
  - Mehiläinen Jyväskylä Occupational Health Services, Jyväskylä
  - Central Finland Hospital District (Perusterveydenhuollon liikelaitos Seututerveyskeskus), Jyväskylä
  - Oma Lääkärisi Tikkakoski, Jyväskylä
  - Oma Lääkärisi Korpilahti, Jyväskylä
  - Sote kuntayhtymä/Perusturvaliikelaitos Saarikka, Saarijärvi

REFERENCES:
- [Derived] Tahkola A, Korhonen P, Kautiainen H, Niiranen T, Mantyselka P. The impact of antihypertensive treatment initiation on health-related quality of life and cardiovascular risk factor levels: a prospective, interventional study. BMC Cardiovasc Disord. 2021 Sep 16;21(1):444. doi: 10.1186/s12872-021-02252-7. PMID 34530733
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Tahkola A, Korhonen P, Kautiainen H, Niiranen T, Mantyselka P. Feasibility of a checklist in treating hypertension in primary care - base line results from a cluster-randomised controlled trial (check and support). BMC Cardiovasc Disord. 2018 Dec 19;18(1):240. doi: 10.1186/s12872-018-0963-5. PMID 30567497